CLINICAL TRIAL: NCT03367637
Title: A Novel mHealth Approach to Assess and Manage Palliative Care Needs for Cancer Patients in Kigali
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Rwanda Palliative Care and Hospice Organization (Unknown); University of California, San Francisco (Other); Cornell Tech (Other); King's College London (Other)
Responsible Party: Principal Investigator, Aparna Parikh, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017P002380
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Cancer Pain
Keywords: Cancer Pain, Palliative care, Mobile Applications, Rwanda
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: We will enroll 80 advanced cancer patients with moderate to severe pain needs (10 per month) with estimated 40% females. Following informed consent, study staff will administer baseline assessments, assess eligibility and obtain consent. Subsequently, eligible consenting patients, will be randomly assigned via computer-generated randomization, to standard palliative care (currently provided at Rwanda Palliative Care and Hospice Organization) or to the new smartphone intervention (with biweekly and SOS symptom assessment and response) plus standard care for 3 months. The probability of being assigned to either group will be equal (50%).
  With 36 patients per group, we will have 85% power to detect a clinically significant difference of 1 point on the pain score [SD=1.4] between the two treatment groups at 3-months with an alpha of 0.05. Based on prior studies and assuming an attrition rate of no more than 10%, we increased our sample size to 40 patients per group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Patients in this arm will receive standard palliative care currently provided at the Rwanda Palliative and Hospice Care Organization (RPCHO).
  Standard care also includes regular follow-up phone calls and home visits by the RPCHO staff, though the timing of these calls is variable and is selected by the discretion of the team. In addition, patients can contact providers on a landline number available during business hours and staffed by an on-call palliative care provider as and when needed.
  Interventions: Other: Standard palliative care
- Intervention (Experimental): Patients in this arm, in addition to the standard palliative care currently provided at the RPCHO, will receive biweekly frequency reminders to fill out the African Palliative Care Outcomes Scale (APCA POS) on the new smart phone based symptom evaluation application on their phones. It is a short symptom assessment questionnaire with responses on 5-point severity scale. In addition to bi-weekly, patients can complete the symptom assessment at any time they feel their symptoms are poorly controlled. The team at RPCHO will be able to track all enrolled patients on a desktop dashboard. Any score of 2 or higher will be flagged. The providers at RPCHO will respond to such patients during business hours via call or text and will advise the patients as indicated or triage to a fellow team member.
  Interventions: Other: Smart Phone based symptom evaluation application

INTERVENTIONS:
Other: Standard palliative care — Standard care includes regular follow-up phone calls and home visits by the RPCHO staff for all advanced cancer patients at RPCHO, though the timing of these calls is variable and is selected by the discretion of the team. In addition, patients can contact providers on a landline number available during business hours and staffed by an on-call palliative care provider as and when needed. For after-hours emergency assistance, patients have the option of contacting the on-call palliative-care physicians for assistance.
  Arms: Standard Care
Other: Smart Phone based symptom evaluation application — In addition to the standard palliative care currently provided at the RPCHO, patients will receive biweekly reminders to fill out the African Palliative Care Outcomes Scale (APCA POS) on the new smartphone application on their phones. It is a short symptom assessment questionnaire with responses on 5-point severity scale. In addition to bi-weekly frequency, patients can complete the symptom assessment at any time they feel their symptoms are poorly controlled. The team at RPCHO will be able to track all enrolled patients on a desktop dashboard. Any score of 2 or higher will be flagged. The providers at RPCHO will respond to such patients during business hours via call or text and will advise the patients as indicated or triage to a fellow team member.
  Arms: Intervention

SUMMARY:
Palliative care is an approach that improves the quality of life of patients and their families facing the problem associated with life-threatening illness such as cancer, through the prevention and relief of suffering by means of early identification and treatment of pain and other physical and psychosocial problems. Despite the rising incidence of cancer, the availability of comprehensive palliative care services across Sub Saharan Africa is extremely limited. The current study will test the efficacy of the newly developed smart phone based symptom evaluation app (application), in improving the management of the palliative care needs of patients with advanced cancer in Rwanda.

RPCHO is the Rwanda Palliative Care and Hospice Organization that provides palliative care services to advanced cancer patients in Rwanda. About 80 patients enrolled under the RPCHO will be enrolled in the current study. Those who agree to take part in the study will be randomly assigned to either a standard care group or intervention group. Patients in both the arms will continue to receive the standard palliative care currently provided at the RPCHO. Additionally, patients in the intervention group will receive new smart-phone application based alerts, bi-weekly, on their mobile phone to fill out the short symptom assessment form. In addition, patients will also be able to complete a symptom assessment at any time they feel that their symptoms are poorly controlled or getting worse. The team at RPCHO will have desktop based dashboard where they will be able to track all patient's information. This will assist them in early identification and response to any worsening symptoms. Patients enrolled in both standard arm and intervention arm, will be asked to make three visits at the RPCHO at baseline, at 6 weeks, at 3 months. During this visits the RPCHO research staff will conduct their physical and psychological assessment.

We hope to find significant improvement in pain score, other symptoms and quality of life, as measured by standard validated scores, for patients enrolled under the intervention arm (using the smart phone app) as compared to standard care arm at 6 weeks and at 3 months. Thus we hope to demonstrate that the new smartphone-based app can be successfully used for both the assessment and management of pain and other symptoms and providing palliative care services for advanced cancer patients in low and middle income countries.

DETAILED DESCRIPTION:
The aim of the study is to conduct a preliminary efficacy study of a smartphone based symptom management app in a small pilot randomized controlled trial (RCT).

We will enroll 80 advanced cancer patients with moderate to severe pain needs (10 per month) with estimated 40% females. Following informed consent, study staff will administer baseline assessments. Subsequently, patients will be randomly assigned via computer-generated randomization, to standard care or to the smartphone intervention plus standard care for 3 months.

In the intervention arm participants will receive twice-weekly smartphone reminders to fill out the APCA POS on their phones. When prompted, participants will be asked to respond to the questions with a numerical value on the 5-point scale. Responses of 2 or higher will be highlighted on the provider's dashboard and identified, as "needs follow-up." Providers will respond to the "needs follow-up" messages (via call or text) and will advise the patients as indicated during business hours. The APCA POS score and any adjustment in medications and advice given will be noted in the medical record and the study software as outlined.

In the standard Care arm patients will get the current palliative care provided at the RPCHO. This standard care includes regular follow-up phone calls and home visits, though the timing of these calls is variable and is selected by the discretion of the team. Patients can also contact RPCHO providers on a landline number available during business hours and staffed by an on-call palliative care provider.

For after-hours emergency assistance, patients in both study arms will still have the option of contacting the on-call palliative-care physicians for assistance, as they do now.

A trained study interviewer, who is blinded to patient assignment, will administer the baseline, 6-week and 3-month assessments for patients in both arms. In the baseline assessment information on patient and disease characteristic (age, sex, marital status, diagnosis, place of care, performance status) and family context (living situation) will be collected. On follow-up visits at 6 week and 3 month, patient's physical and psychosocial assessment will be done through expanded APCA POS (African Palliative Care Outcome Scale). APCA POS have been previously validated in the African setting. The APCA POS includes ten questions in total, two focused on physical symptoms including pain and assessment of general symptoms, five focused on psychosocial needs and three questions focused on the care-giver perspective of needs. Because our study is focused on the tracking and monitoring of physical symptoms of patients, three additional questions from the Palliative Outcomes Scale - Symptom List (POS-S) are added to the APCA POS which include shortness of breath, nausea and vomiting, fatigue and constipation.

The assessment will be completed via paper and pencil and entered by the project coordinator into a password-protected, de-identified database, using double data entry, and uploaded to an encrypted, password protected, shared database which the PIs will be responsible for maintaining. All information pertaining to smartphone messages, including patient and provider responses will also be uploaded into the encrypted password-protected software maintained by Cornell Tech.

Primary outcome for the study is difference in pain score as measured by the expanded APCA POS in two arms. Secondary outcomes are difference in other symptoms and quality of life (QOL) scores from the remaining portion of the expanded APCA POS individually and as composite score between the two arms. We will examine the efficacy of the app to improve these outcomes at 6 weeks and 3 months, adjusting for baseline scores with intension-to-treat analysis. These data will help us determine effect size used for sample size calculation of a future large scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Diagnosed with advanced cancer and in moderate or severe pain, as defined by use of World Health Organization (WHO) as requiring step 2 drugs (Tramadol or Codeine) or WHO step 3 drugs (narcotics other than Codeine) to manage their pain.
* Eligible patients or their primary care giver must have a smartphone and/or have a family member that lives at home with a smartphone; and

Exclusion Criteria:

* Projected life expectancy of <3 months at the time of enrollment, to be estimated by their healthcare provider
* Patients enrolled in the smartphone application development phases (earlier than RCT) of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Difference in pain score as measured by the expanded African Palliative Care Outcomes Scale (APCA POS) | 6 weeks, 3 months
  Pain score will be assessed on a scale 1(no pain)-5 (worst/overwhelming pain) in both arms and the mean difference in pain score between two arms will be calculated.

SECONDARY OUTCOMES:
Difference in other symptoms and quality of life (QOL) scores from the remaining portion of the expanded APCA POS individually and as composite score. | 6 weeks, 3 months
  Physical symptoms, psychosocial needs, and caregiver's perspective of patient need will be assessed on a scale 1 (better)-5(worse) [except for questions 4 to 9 in original APCA POS which are scaled 1(worse) to 5(better)] in both arms and the mean difference in the scores between two arms will be calculated individually and as a composite QOL score. The composite QOL will be generated by totaling scores from each question, and the production of a rating against a range of scores from 0-50 for patients (0-35 for the 7 patient related questions in the original APCA POS and 0-15 for additional 3 symptom related questions we added from POS-S) and 0-15 for family members/caretakers. To ensure that all scores are correctly directed (i.e. the lower the score the better the outcome against an item, the higher the score, the more severe the outcome), we will reverse the scores for questions 4-9 in the original APCA-POS for the purpose of data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Parikh, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Rwanda Palliative Care and Hospice Organization (RPCHO), Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ntizimira CR, Nkurikiyimfura JL, Mukeshimana O, Ngizwenayo S, Mukasahaha D, Clancy C. Palliative care in Africa: a global challenge. Ecancermedicalscience. 2014 Dec 11;8:493. doi: 10.3332/ecancer.2014.493. eCollection 2014. PMID 25624874
- [Background] Sepulveda C, Habiyambere V, Amandua J, Borok M, Kikule E, Mudanga B, Ngoma T, Solomon B. Quality care at the end of life in Africa. BMJ. 2003 Jul 26;327(7408):209-13. doi: 10.1136/bmj.327.7408.209. PMID 12881267
- [Background] Clark D, Wright M, Hunt J, Lynch T. Hospice and palliative care development in Africa: a multi-method review of services and experiences. J Pain Symptom Manage. 2007 Jun;33(6):698-710. doi: 10.1016/j.jpainsymman.2006.09.033. PMID 17531910
- [Background] Harding R, Selman L, Agupio G, Dinat N, Downing J, Gwyther L, Mashao T, Mmoledi K, Moll T, Sebuyira LM, Panjatovic B, Higginson IJ. Validation of a core outcome measure for palliative care in Africa: the APCA African Palliative Outcome Scale. Health Qual Life Outcomes. 2010 Jan 25;8:10. doi: 10.1186/1477-7525-8-10. PMID 20100332
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Kroenke K, Krebs EE, Wu J, Yu Z, Chumbler NR, Bair MJ. Telecare collaborative management of chronic pain in primary care: a randomized clinical trial. JAMA. 2014 Jul 16;312(3):240-8. doi: 10.1001/jama.2014.7689. PMID 25027139
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Agboola S, Kamdar M, Flanagan C, Searl M, Traeger L, Kvedar J, Jethwani K. Pain management in cancer patients using a mobile app: study design of a randomized controlled trial. JMIR Res Protoc. 2014 Dec 12;3(4):e76. doi: 10.2196/resprot.3957. PMID 25500281